CLINICAL TRIAL: NCT00698061
Title: A Study to Compare the Immunogenicity and Safety of GSK Biologicals Adjuvanted HBV Vaccine to Engerix™-B, in a Non-responder Population ≥ 15 Years of Age, When Administered Intramuscularly, According to a 0, 1, 2, 12 Month Schedule
Brief Title: Immunogenicity and Safety of an Adjuvanted HBV Vaccine Compared to Engerix™-B, in a Non-responder Population ≥ 15y
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 208129/033; 208129/038 (Other: GSK)
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Adjuvanted vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 3-dose primary vaccination and booster vaccination by intramuscular injection
  Arms: Group A
Biological: Engerix™-B — 3-dose primary vaccination and booster vaccination by intramuscular injection
  Arms: Group B

SUMMARY:
Subjects who had not responded to previous hepatitis B vaccination were vaccinated with either the adjuvanted HBV-MPL vaccine or Engerix™-B vaccine according to a three-dose vaccination schedule (0, 1, 2 months) and boosted at Month 12 as per their group allocation. The immunogenicity and safety of the HBV-MPL vaccine were compared with the control vaccine, Engerix™-B.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham.

ELIGIBILITY:
Inclusion Criteria:

At study entry:

* A male or female ≥ 15 years of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the subject.
* Documented non-response to previous hepatitis B vaccination within 6 months after having received a full vaccination course (i.e. ≥ 3 doses of a hepatitis B vaccine)
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or use adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination.

Before booster dose at month 12:

* Additional written informed consent covering the booster administration and blood samples at months 12 and 13 must be obtained from the subject.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or use adequate contraceptive precautions for one month prior to and up to two months after the administration of the booster dose

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Known exposure to hepatitis B within 6 weeks.
* History of hepatitis B infection.
* Confirmed human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease/reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration/ administration during the study period.
* Pregnant or lactating female.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 1999-11; Primary Completion 2000-09 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | Months 1, 2 and 3

SECONDARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general signs and symptoms | During a 4 day follow-up period after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited signs and symptoms | During a 30 day follow-up period after vaccination
Occurrence, intensity and relationship to vaccination of serious adverse events (SAEs) | During the study period, up to and including 6 months post-vaccination
Anti-HBs antibody concentrations in all subjects | Months 1, 2, 3, 12 and 13

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199